CLINICAL TRIAL: NCT05484284
Title: Can Two-stage Primary Total Knee Arthroplasty With Low-dose Antibiotics Effectively Treat Septic Arthritis of the Native Knee Joint?
Brief Title: Two-stage Arthroplasty for the Septic Arthritis of the Native Knee Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0292
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Septic Arthritis
MeSH Terms: conditions — Arthritis, Infectious | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All the patients (Experimental): patients received two-stage primary total knee arthroplasty with low-dose antibiotics
  Interventions: Procedure: two-stage primary total knee arthroplasty with low-dose antibiotics

INTERVENTIONS:
Procedure: two-stage primary total knee arthroplasty with low-dose antibiotics — Briefly, investigators completely debrided all necrotic soft tissue in the first stage of the operation. The surgical site was flushed twice with hydrogen peroxide, iodine, and saline solutions. Then, the antibiotic-loaded cement spacer was inserted. After surgery, a 10-day course of intravenous organism-specific antibiotics or vancomycin was administered, followed by oral antibiotic therapy. Second-stage reimplantation was performed once there was no sign of infection. The spacer was removed and the new prosthesis was implanted without the use of antibiotic-containing bone cement.

SUMMARY:
Septic arthritis (SA) of the native knee joint is rare but difficult to manage. Open or arthroscopic debridement is currently the most widely used approach. The problem is that there is a 71% and 50% chance of requiring revision surgery, respectively. Patients with recurrent sepsis may require arthrodesis or amputation, which would result in severe functional loss. Therefore, there is an urgent need to find more effective surgical procedures. Investigators developed a two-stage exchange with low-dose antibiotics for the treatment of SA and evaluated its efficacy.

DETAILED DESCRIPTION:
Septic arthritis (SA) of the native knee joint is a rare but highly disabling disease. Epidemiologic studies have documented an incidence of 0.9 per 100,000. The treatment is challenging and the ideal treatment strategy is not well established. Over the past decades, open or arthroscopic debridement with systemic antibiotic therapy is the most widely used approach. However, a recent study has shown that these two methods have a failure rate as high as 50%-71%. Patients with recurrent sepsis may require arthrodesis or amputation, which would result in severe functional loss. Therefore, there is an urgent need to find more effective surgical procedures.

A few reports proposed two-stage exchange to address SA and showed satisfying clinical outcomes. Orthopedic surgeons removed the infected soft and bone tissue during the first operation and then implant antibiotic-loaded bone cement spacer. Once the infection had been addressed, a new prosthesis was inserted in a second operation. This approach could greatly boost the success rate to over 95%. However, the issue is that high-dose antibiotics bone cement may cause life-threatening complications such as acute kidney injury and drug-induced immune hemolytic anemia. Therefore, investigators developed a two-stage exchange with low-dose antibiotics for the treatment of SA.

Investigators summarized and analyzed the treatment processes and performed laboratory, imaging, and functional evaluations after treatment. The purpose was to introduce a new treatment regimen for SA and evaluate the technical points of the regimen, and prognosis over medium-term follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with SA based on one or more of the following: clinical presentations (fever, joint pain, restricted mobility, swelling and redness, and/or a discharging sinus communicating with the joint); elevated inflammation markers; evidence of infection on images; purulence in the joint, and positive frozen section or cultures
* Without infections at other sites
* Without venous thrombosis of the lower limbs
* American society of Anesthesiologists (ASA) physical status classification was either 1 or 2
* With complete data for the main indicators (routine blood test results, C-reactive protein level, erythrocyte sedimentation rate, X-ray and/or MRI scans of the surgical site, and the Knee Society Function scores).

Exclusion Criteria:

* Patients (<60 yrs) without progression to advanced osteoarthritis
* In poor general condition who could not tolerate surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Surgical success rate | two years postoperatively
  The clearance rate of infection
Surgical success rate | three years postoperatively
  The clearance rate of infection
Surgical success rate | four years postoperatively
  The clearance rate of infection
Surgical success rate | five years postoperatively
  The clearance rate of infection
Surgical success rate | six years postoperatively
  The clearance rate of infection
Surgical success rate | seven years postoperatively
  The clearance rate of infection
Surgical success rate | eight years postoperatively
  The clearance rate of infection

SECONDARY OUTCOMES:
change from baseline in knee joint function | baseline, 1 month, 2 month, 3 month, 6 month, and yearly postoperatively
  record Knee Society Function scores (0-100), the higher the score, the better the function

CONTACTS AND LOCATIONS:
Overall Officials: Lan Tang, MD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ross JJ. Septic Arthritis of Native Joints. Infect Dis Clin North Am. 2017 Jun;31(2):203-218. doi: 10.1016/j.idc.2017.01.001. Epub 2017 Mar 30. PMID 28366221
- [Background] Mathews CJ, Weston VC, Jones A, Field M, Coakley G. Bacterial septic arthritis in adults. Lancet. 2010 Mar 6;375(9717):846-55. doi: 10.1016/S0140-6736(09)61595-6. PMID 20206778